CLINICAL TRIAL: NCT00003153
Title: Phase II Study of Salvage Cellular Immunotherapy for Patients With Persistent or Recurrent Multiple Myeloma After Allogeneic Bone Marrow Transplantation From an HLA-Matched Sibling Donor
Brief Title: Biological Therapy in Treating Patients With Multiple Myeloma That Has Recurred Following Bone Marrow Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065938; ECOG-E1A97
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes

SUMMARY:
RATIONALE: White blood cells from donors may be able to kill cancer cells in patients with multiple myeloma that has recurred following bone marrow transplantation.

PURPOSE: This phase II trial is studying how well giving donor white blood cells works in treating patients with recurrent multiple myeloma who have undergone bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the response rate of patients with recurrent multiple myeloma after an allogeneic marrow transplant from a genotypically HLA identical sibling donor treated with donor lymphocyte infusions as salvage therapy .
* Evaluate the safety and toxicity of this treatment when used as salvage therapy in these patients.

OUTLINE: Patients receive initial cell dose of donor lymphocytes (CD3+ cells) IV over 15-30 minutes. Patients with rapidly progressive disease may skip the initial cell dose and proceed directly to dose escalation to receive CD3+ cells at a higher cell dose. Patients who achieve complete response to the initial treatment may receive up to 2 additional courses of escalating doses of CD3+ cells 8-12 weeks apart in the absence of unacceptable toxicity. Patients are evaluated at 4 and 8 weeks after each infusion. Patients with disease progression at 8 weeks are retreated at that time. Patients who achieve partial response or stable disease at 8 weeks are re-evaluated at 12 weeks and may then be retreated.

Patients are followed every 2 weeks for 3 months, once a month for 9 months, and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 22 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or persistent multiple myeloma at least 6 months following allogeneic bone marrow transplantation (BMT) from an HLA identical sibling
* Must meet one of following criteria to be considered persistent, recurrent, or progressive disease:

  * Residual detectable disease 6-12 months after BMT, as determined by the M protein level or bone marrow involvement, without further evidence of clinical or laboratory improvement on 2 consecutive measurements 4 weeks apart
  * Complete response not achieved 12 or more months after BMT and there is no evidence of progressive improvement
  * At least 25% increase of serum paraprotein (greater than 1.0 g/dL) as measured on two occasions or a 50% increase in urinary light chain excretion (greater than 150 mg/day) as measured on 2 occasions
  * A 10% increase in plasma cells in the bone marrow
* Disease in complete response but with recurrence of M protein and 10% point increase in myeloma cells in the marrow allowed
* No lytic lesions alone or new soft tissue plasmacytoma as sole evidence of progression

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 4 weeks

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 times upper limit of normal

Renal:

* Not specified

Other:

* No active infection
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Must have received prior allogeneic bone marrow transplantation from an HLA A;B;DR genotypically matched sibling donor
* No concurrent interferon therapy for relapsed disease

Chemotherapy:

* At least 4 weeks since cyclosporine, methotrexate, azathioprine, or other graft versus host disease (GVHD) prophylaxis/treatment without evidence of flare of GVHD
* At least 4 weeks since prior chemotherapy for relapsed disease

Endocrine therapy:

* Must be receiving a dose no greater than 0.25 mg/kg prednisone for at least 4 weeks prior to registration without flare of GVHD
* No prior prednisone dose greater than 0.25 mg/kg in the past 4 weeks
* Must receive concurrent prednisone of a dose no greater than 0.25 mg/kg
* Concurrent corticosteroids allowed

Radiotherapy:

* Concurrent palliative radiotherapy allowed if evidence of other evaluable disease other than irradiated bony sites

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 1998-07-22 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Vesole DH, Zhang L, Flomenberg N, Greipp PR, Lazarus HM, Huff CA; ECOG Myeloma and BMT Committees. A Phase II trial of autologous stem cell transplantation followed by mini-allogeneic stem cell transplantation for the treatment of multiple myeloma: an analysis of Eastern Cooperative Oncology Group ECOG E4A98 and E1A97. Biol Blood Marrow Transplant. 2009 Jan;15(1):83-91. doi: 10.1016/j.bbmt.2008.10.030. PMID 19135946